CLINICAL TRIAL: NCT03270722
Title: Use of FLIP Topography to Evaluate Esophageal Symptoms in Patients With Scleroderma
Brief Title: Functional Luminal Imaging Probe (FLIP) Topography Use in Patients With Scleroderma and Trouble Swallowing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We did not enroll any patients for logistic reasons.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Zikos, Fellow in Gastroenterology, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-42435
Record Dates: First submitted 2017-08-18; First posted 2017-09-01 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Scleroderma; Dysphagia; GERD - Gastro-Esophageal Reflux Disease
MeSH Terms: conditions — Scleroderma, Diffuse; Deglutition Disorders; Gastroesophageal Reflux | interventions — Gastroscopy; Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- patients with scleroderma and trouble swallowing (Experimental)
  Interventions: Device: FLIP topography; Procedure: Upper Endoscopy
- patients with scleroderma but no trouble swallowing (Experimental)
  Interventions: Device: FLIP topography; Procedure: Upper Endoscopy
- patients without scleroderma undergoing endoscopy (Active Comparator)
  Interventions: Device: FLIP topography; Procedure: Upper Endoscopy

INTERVENTIONS:
Device: FLIP topography — During upper endoscopy, the FLIP topography balloon will be advanced into the esophagus and inflated, providing additional information about the distensibility of the esophagus. This generally takes about 5 extra minutes and no complications have been reported. Theoretical complications include bleeding, infection, risk with extra anesthesia time, and putting a hole in the esophagus.
Procedure: Upper Endoscopy — A standard upper endoscopy will also be done in all patients. A small scope will be passed via the mouth to examine the esophagus, stomach, and first part of the small intestine. The risks of this procedure include the risks associated with anesthesia, a small risk of bleeding, infection, and a very small risk of putting a hole in the gastrointestinal tract.
  Other Names: EGD (esophagogastroduodenoscopy)

SUMMARY:
FLIP topography has been FDA cleared to evaluate a variety of esophageal conditions, but has never been evaluated in patients with scleroderma. The investigators hope to evaluate this technology in patients who have scleroderma and various esophageal symptoms, and compare to non-scleroderma patients.

DETAILED DESCRIPTION:
In patients with treatment refractory reflux disease, dysphagia (trouble swallowing) or other symptoms possibly attributed to the esophagus, the standard protocol is generally to first do an upper endoscopy to evaluate for abnormalities. If this is normal the next step is often to do esophageal manometry to measure esophageal muscle contractions, along with a Ph/impedance study in certain clinical situations. If these are normal, then the the disorder is thought to be functional (no clear biological pathology). However, it is believed that FLIP (Functional Luminal Imaging Probe) technology may pick up additional disorders of the esophagus missed by standard esophageal manometry, leading to different treatments in certain cases. Additionally, FLIP technology offers a different approach to classifying motility disorders of the esophagus.

FLIP is a technology that measures distensibility and diameter of the esophagus during endoscopy by inflating a balloon in the esophagus. It has previously been used to aid in the diagnosis and provide more information regarding gastroesophageal reflux disease, achalasia, and eosinophilic esophagitis. It has also been used pre and post fundoplication and myotomy to assess adequacy of these procedure.

More recently a group at northwestern has developed a modification of this procedure called FLIP topography. The basic principles are the same, but this technique measures the reaction of the esophagus to distension, providing additional information.

A recent study of FLIP topography looked at 145 patients referred for dysphagia (trouble swallowing). All patients had both standard manometry and FLIP topography. 25% of patients in the study had a normal manometry, offering no measurable explanation of their symptoms. Of these patients, half had an abnormal FLIP topography, and additional treatments were offered in certain situations.

FLIP topography has also been evaluated in patients with eosinophilic esophagitis, though numbers are small.

Currently, the FLIP topography device has been FDA cleared for esophageal distensibility testing. It has never been evaluated specifically in patients with scleroderma.

ELIGIBILITY:
Inclusion Criteria:

* Must have a clinical indication for upper endoscopy (recruiting patients both with scleroderma and without)

Exclusion Criteria:

* not healthy enough to undergo an upper endoscopy
* mass, stricture, ring, or web present on upper endoscopy
* history of esophageal cancer
* history of esophageal surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
FLIP topography pattern | Will be analyzed directly after the procedure for an individual patient within 2 weeks. Comparisons within and between the 3 groups will be done at the conclusion of the study (once 60 total patients have been recruited).
  This is the readout or topographic map that is generated from the FLIP topography diagnostic procedure. We will look to see if we can make additional diagnoses not made by other clinical testing, to see if the diagnoses made by FLIP topography match with other diagnostic testing, and identify new FLIP topography patterns in patients with scleroderma not seen before.

SECONDARY OUTCOMES:
Change in medical management | Recommendations will be made directly after the procedure. Chart reviews at 6 months will also occur to monitor implementation of medical recommendations.
  The investigators will look to see if FLIP topography lead to the recommendation of additional medicines and/or surgeries/procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Healthcare, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No